CLINICAL TRIAL: NCT00635843
Title: "A Prospective, Randomized Controlled Clinical Investigation of MAVERICK™ Total Disc Replacement in Patients With Degenerative Disc Disease"
Brief Title: MAVERICK™ Total Disc Replacement- Pivotal Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-08
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Diseases
Keywords: Lumbar degenerative disc disease at one level from L4-S1
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAVERICK™ Disc (Experimental)
  Interventions: Device: MAVERICK™ Disc
- Fusion (Active Comparator)
  Interventions: Device: LT-CAGE® Lumbar Tapered Fusion Device and INFUSE® Bone Graft

INTERVENTIONS:
Device: MAVERICK™ Disc — The MAVERICK™ disc is a spinal arthroplasty system and is intended to replace a damaged disc in the lumbar spine. It is a permanent implant used to maintain motion at the treated level and is inserted using an anterior surgical approach.
  Other Names: MAVERICK™
  Arms: MAVERICK™ Disc
Device: LT-CAGE® Lumbar Tapered Fusion Device and INFUSE® Bone Graft — The control is the treatment with LT-CAGE® Lumbar Tapered Fusion Device and INFUSE® Bone Graft. It is commercially available for anterior lumbar spine interbody fusion procedures.
  Other Names: Fusion
  Arms: Fusion

SUMMARY:
The purpose of this clinical trial is to assess the safety and effectiveness of the MAVERICK™ Total Disc Replacement as a method of treating patients with lumbar degenerative disc disease at one level from L4-S1, with overall success being the primary endpoint of the clinical trial. The primary objective is to show non-inferiority of the investigational device to the control treatment. If non-inferiority is established, superiority will be examined.

DETAILED DESCRIPTION:
For this clinical trial, there are two treatment groups, i.e., investigational patients who receive the MAVERICK™ Total Disc Replacement and control patients who receive the anterior lumbar interbody fusion procedure with INFUSE® Bone Graft/LT-CAGE® Lumbar Tapered Fusion Device. Each investigational site will enroll patients in a 2:1 investigational:control treatment randomization scheme.

ELIGIBILITY:
Inclusion Criteria:

* Has DDD as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history
* Has 1 or more of the following documented by CT, MRI, or plain x-rays: modic changes, high intensity zones in the annulus, loss of disc height, decreased hydration of the disc
* Has documented annular pathology
* Has single-level symptomatic degenerative involvement from L4-S1 requiring surgical treatment
* Has intact facet joints at the involved vertebral levels documented by CT and/or MRI
* Has preop Oswestry score≥30
* Has preop back pain score ≥20
* Age 18 to 70 yrs who are skeletally, mature, inclusive
* Has not responded to non-operative treatment for 6 mos
* If child-bearing potential, patient is non-pregnant, non-nursing, and agrees not to become pregnant for 1 yr after surgery
* Is willing and able to comply with the study plan and sign the Patient Informed Consent Form

Exclusion Criteria:

* Has primary diagnosis of a spinal disorder other than DDD at involved level
* Had previous posterior lumbar spinal fusion surgical procedure at involved level
* Had prior posterior lumbar surgery resulting in significant muscle/ligament morbidity, not including facet saving techniques
* Had previous anterior lumbar spinal surgery at involved level
* Requires spinal fusion and/or arthroplasty at more than 1 lumbar level
* Has severe pathology of facet joints of involved vertebral bodies
* Has any posterior element insufficiency
* Has spondylolisthesis
* Has spinal canal stenosis
* Has rotatory scoliosis at involved level
* Level treated has fractures secondary to trauma
* Has any of the following that may be associated with a diagnosis of osteoporosis (if Yes, a DEXA Scan is required): Postmenopausal Non-Black female over 60 yrs of age and weighs less than 140 pounds; Postmenopausal female that has sustained a non-traumatic hip, spine or wrist fracture; Male over the age of 60 that has sustained a non-traumatic hip or spine fracture. If level of BMD is -3.5 or lower or -2.5 or lower with vertebral crush fracture, the patient is excluded
* Has fever (temp > 101°F oral) at time of surgery
* Has a condition that requires postop medications that interfere with fusion, such as steroids or prolonged use of non-steroidal anti-inflammatory drugs, excluding routine perioperative, non-steroidal anti-inflammatory drugs. Does not include low dose aspirin for prophylactic anticoagulation
* Has overt or active bacterial infection, either local or systemic and/or potential for bacteremia
* Has presence or prior history of malignancy (except for basal cell carcinoma of skin)
* Has documented metal allergy, titanium alloy intolerance or cobalt-chrome-molybdenum alloy
* Is mentally incompetent. If questionable, obtain psych consult
* Has a Waddell Signs of Inorganic Behavior score of 3 or greater
* Has chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease
* Is prisoner
* Is pregnant
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse
* Has received drugs that may interfere with bone metabolism within 2 weeks prior to the surgery date, excluding routine perioperative, non-steroidal anti-inflammatory drugs
* Has history of autoimmune disease
* Has history of exposure to injectable collagen implants
* Has history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen
* Has received treatment with an investigational therapy within 30 days prior to implantation surgery or treatment is planned during 24 months following the implantation surgery
* Has received any previous exposure to any/all BMP's of either human or animal extraction
* Has history of allergy to bovine products or a history of anaphylaxis
* Has history of any endocrine or metabolic disorder known to affect osteogenesis
* Has any disease that would preclude accurate clinical evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2003-04; Primary Completion 2006-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall Success | 24 Months
  A patient will be considered an overall success if all of the following conditions are met:
  1. pain/disability(Oswestry)success;
  2. neurological status success;
  3. disc height success;
  4. no serious adverse event classified as "implant associated" or "implant/surgical procedure associated";
  5. no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
Pain/Disability Status | 24 Months
  The self-administered Oswestry Low Back pain Disability Questionnaire will be used. Success will be defined as pain/disability improvement postoperatively according to the following definition:
  Preoperative Score - Postoperative Score >= 15
Neurological Status | 24 months
  Neurological status will be evaluated preoperatively and postoperatively. Neurological status is based on four types of measurements (sections): motor, sensory, reflexes, and straight leg raise. Each of the categories is comprised of a number of elements. Postoperative evaluations on each element on the Neurological status case report form will be compared to the preoperative evaluations. Success will be defined as maintenance or improvement in each element for the time period evaluated.
Disc Height Measurement | 24 months
  Disc height will be measured postoperatively at each visit and compared to the measurement at 6 weeks postoperatively. Disc height success is based on either the anterior or posterior measurements meeting the following criterion:
  Postoperative Disc Height- 6 Week Postoperative Disc Height >= -2mm
General Health Status | 24 months
  The Medical Outcomes Study 36-item Short Form Health Survey (SF-36) will be used to assess general health status. The SF-36 results can be summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). Success will be defined as a maintenance or improvement in status postoperatively as compared to the preoperative condition. To be classified as a success, the following criteria must be met:
  PCSPostop - PCSPreop >= 0; MCSPostop - MCSPreop >= 0
Back Pain | 24 months
  Numerical rating scales will be used to evaluate pain intensity and duration. The pain score (0 min, 20 Max) is derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and duration scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Success for back and leg pain is described as follows:
  Preoperative Score - Postoperative Score >0
Leg Pain | 24 months
  Numerical rating scales will be used to evaluate pain intensity and duration. The pain score (0 min, 20 Max) is derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and duration scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Success for back and leg pain is described as follows:
  Preoperative Score - Postoperative Score >0
Patient Satisfaction | 24 months
Patient Global Perceived Effect | 24 months
Operative Time | At the time of operation
Blood Loss | At the time of operation
Number of Hospital Days | At the time of discharge

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - The Spine Center at TOC, Huntsville, Alabama
  - Spine Care Medical Group, Daly City, California
  - Little Company of Mary Hospital, Los Angeles, California
  - Newport Orthopedic Institute, Newport Beach, California
  - Orthopaedic Specialty Institute, Orange, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - Rocky Mountain Associates in Orthopaedic Medicine, Loveland, Colorado
  - Orthopaedic & Sports Medicine Center, Trumbull, Connecticut
  - First State Orthopaedics, P.A., Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - The B.A.C.K. Center, Melbourne, Florida
  - Hughston Clinic, Columbus, Georgia
  - Spine Institute of Idaho, Meridian, Idaho
  - Northwestern Orthopedic Institute, Chicago, Illinois
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Orthopedics of Indianapolis, Indianapolis, Indiana
  - Institute for Low Back & Neck Care, Minneapolis, Minnesota
  - Orthopedic Center of St. Louis, Chesterfield, Missouri
  - Nebraska Spine Center, LLC, Omaha, Nebraska
  - New Hampshire Spine Institute, Bedford, New Hampshire
  - Hospital for Special Surgery, New York, New York
  - Spine Carolina, Asheville, North Carolina
  - Oklahoma Sports Science & Ortho, Oklahoma City, Oklahoma
  - Southeastern Spine Institute, Mt. Pleasant, South Carolina
  - Central Texas Spine, Austin, Texas
  - The Center for Spine Care, Dallas, Texas
  - Advanced Neurosurgical Center, El Paso, Texas
  - Virginia Spine Institute, Reston, Virginia
  - Neurosurgical Associates, PC, Richmond, Virginia
  - Inland Neurosurgery and Spine Associates, PS, Spokane, Washington
  - University of Wisconsin Orthopedic Department, Madison, Wisconsin

REFERENCES:
- [Derived] Gornet MF, Burkus JK, Dryer RF, Peloza JH, Schranck FW, Copay AG. Lumbar disc arthroplasty versus anterior lumbar interbody fusion: 5-year outcomes for patients in the Maverick disc investigational device exemption study. J Neurosurg Spine. 2019 May 17;31(3):347-356. doi: 10.3171/2019.2.SPINE181037. Print 2019 Sep 1. PMID 31100723
- [Derived] Burkus JK, Dryer RF, Peloza JH. Retrograde ejaculation following single-level anterior lumbar surgery with or without recombinant human bone morphogenetic protein-2 in 5 randomized controlled trials: clinical article. J Neurosurg Spine. 2013 Feb;18(2):112-21. doi: 10.3171/2012.10.SPINE11908. Epub 2012 Nov 30. PMID 23199378